CLINICAL TRIAL: NCT04171115
Title: A Phase 1, Randomized, Double-Blind, Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of a Single IM Dose of G03-52-01 vs Placebo in Adult Subjects
Brief Title: Study to Evaluate Safety and PK of a Single IM Dose of G03-52-01 vs Placebo in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: G03-52-01.001
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: botulinum toxin; botulism
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Intervention Model Description: dose escalation trial of four dose cohorts of 10 subjects (A: 10mg, B: 25mg, C: 50mg, D: 100 mg)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10mg of G03-52-01 (Experimental): 8 subjects randomized to 10 mg of G03-52-01 and 2 subjects randomized to placebo
  Interventions: Drug: G03-52-01; Drug: Placebo
- 25mg of G03-52-01 (Experimental): 8 subjects randomized to 25 mg of G03-52-01 and 2 subjects randomized to placebo
  Interventions: Drug: G03-52-01; Drug: Placebo
- 50 mg of G03-52-01 (Experimental): 8 subjects randomized to 50 mg of G03-52-01 and 2 subjects randomized to placebo
  Interventions: Drug: G03-52-01; Drug: Placebo
- 100 mg of G03-52-01 (Experimental): 8 subjects randomized to 100 mg of G03-52-01 and 2 subjects randomized to placebo
  Interventions: Drug: G03-52-01; Drug: Placebo

INTERVENTIONS:
Drug: G03-52-01 — G03-52-01 administered intramuscularly
Drug: Placebo — Placebo administered intramuscularly

SUMMARY:
A Phase 1, randomized, double-blind, placebo-controlled dose escalation trial of four dose cohorts of 10 subjects (1: 10mg, 2: 25mg, 3: 50mg, 4: 100mg).

DETAILED DESCRIPTION:
A Phase 1, randomized, double-blind, placebo-controlled dose escalation trial of four dose cohorts of 10 subjects (1: 10mg, 2: 25mg, 3: 50mg, 4: 100mg). Dose escalation will not occur until safety data through Day 8 is reviewed by the Safety Review Committee (SRC). The study will consist of a twenty-eight day screening period, 12-hour clinic stay, and 120-day (Cohorts 1-3) or 180-day (Cohort 4) outpatient follow-up. The primary objective of this study is to assess the safety and tolerability of escalating doses of G03-52-01 administered intramuscularly (IM) in healthy adult subjects. The secondary objectives are to evaluate the pharmacokinetics (PK) and immunogenicity of escalating IM doses of G03-52-01.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood and signed
2. Healthy male or healthy, non-pregnant, non-lactating female
3. Willingness to comply and be available for all protocol procedures
4. Between 18 and 45 years of age on the day of IM injection
5. Body Mass Index (BMI) of ≥18.5 and ≤35 kg/m2
6. If the subject is female and of childbearing potential, she has a negative serum pregnancy test at screening and negative urine test within 24 hours prior to IM injection

   • Note: A woman is considered of childbearing potential unless post-menopausal (≥ 1 year without menses) or surgically sterilized via bilateral oophorectomy, or hysterectomy or bilateral tubal ligation or successful Essure placement with documented confirmation test at least 3 months after the procedure.
7. If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use acceptable contraception during participation in the study

   • Note: Acceptable contraception methods are restricted to effective devices (Intrauterine Contraceptive Devices)
8. The hemoglobin, platelet count, white blood cell count and absolute neutrophil count are not below the LLN and ≤ULN x 10%

   • Abnormalities in mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV), and nucleated red blood cell count (NRBC CT), which are included in a complete blood count with differential, will not be exclusions.
9. The urine dipstick results on protein, glucose and blood are negative or trace

   * Note: Menstruating females failing inclusion criteria due to a positive blood on urine dipstick may be retested following cessation of menses.
   * Note: When a urine dipstick is more than trace positive for blood (whether a menstruating female or other subjects), that subject would not be excluded if the urine microscopic exam shows <5 rbcs/hpf.
10. Chemistry screening laboratory tests as outlined in Section 7.5.1.4 are in the normal reference range

    * Note: The following exceptions to laboratory normal reference ranges are allowed: Creatinine, Blood Urea Nitrogen (BUN), total bilirubin, AST, ALT, lipase, amylase, Prothrombin Time (PT), Partial Thromboplastin Time (PTT) below the lower limit of normal (LLN); CK less than 400U/L; Glucose, potassium, total protein, and alkaline phosphatase with a toxicity grade of 1 is allowable; albumin above the upper limit of normal (ULN).
    * Laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to laboratory error may be repeated once.
11. The urine drug screen is negative
12. Breathalyzer test is negative
13. Available for follow-up for the duration of the study
14. Agrees not to participate in vigorous activity 72 hours prior to dosing through day 15 post dosing

Exclusion Criteria:

1. History of a chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject.

   • Note: Chronic medical conditions include but not limited to diabetes; Asthma requiring use of medication in the year before screening; Autoimmune disorder such as lupus, Wegener's, rheumatoid arthritis, thyroid disease; Coronary artery disease; Chronic hypertension; History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease (except previous asthma which has required no treatment for the past year);
2. History of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins.

   • Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema
3. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds)
4. Clinically significant abnormal electrocardiogram at screening.

   • Note: Clinically significant abnormal ECG results include but not limited to: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator
5. Positive serology results for HIV, HBsAg, or HCV antibodies
6. Febrile illness with temperature ≥38°C within 7 days of dosing
7. Pregnant or breastfeeding
8. Donated blood within 56 days of enrollment
9. Known allergic reactions to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure
10. Treatment with another investigational drug within 28 days of dosing
11. Treatment with a monoclonal antibody within 3 months of enrollment.
12. Receipt of antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
14. Use of H1 antihistamines or beta-blockers within 5 days of dosing
15. Use of any prohibited medication within 28 days prior to study entry or planned use during the study period

    • Note: Prohibited medications include immunosuppressives (except Nonsteroidal Anti-Inflammatory Drugs [NSAIDS]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents; any vaccine (licensed or investigational). Subjects will be eligible to receive any authorized COVID-19 vaccine after they complete Study Day 8
16. Previous exposure to botulinum toxin, receipt of antibodies against botulinum toxin, or previous treatment with equine antitoxin
17. Any previous injection or planned injection within 4 months after enrollment of botulinum toxin for cosmetic reasons, spastic dysphonia, torticollis, or any other reason
18. Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety
19. Plans to enroll or is already enrolled in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period

    • Note: Includes trials that have a study intervention such as a drug, biologic, or device
20. Is a study site employee or staff

    • Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators
21. Systolic blood pressure >140mm Hg or diastolic blood pressure >90 mm Hg
22. Resting hear rate <50 or >100 beats per minute
23. Oral temperature ≥ 38°C (100.4°F)
24. Subjects with NX02 antibody levels present at screening will be excluded from Cohort 4.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Key, MD, Principal Investigator — ICON Early Phase Services, LLC
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10mg of G03-52-01: 8 subjects randomized to 10 mg of G03-52-01
  G03-52-01: G03-52-01 administered intramuscularly
- 25mg of G03-52-01: 8 subjects randomized to 25 mg of G03-52-01
  G03-52-01: G03-52-01 administered intramuscularly
- 50 mg of G03-52-01: 8 subjects randomized to 50 mg of G03-52-01
  G03-52-01: G03-52-01 administered intramuscularly
- 100 mg of G03-52-01: 8 subjects randomized to 100 mg of G03-52-01
  G03-52-01: G03-52-01 administered intramuscularly
- Pooled Placebo: 2 subjects randomized to placebo in each of the 4 cohorts/dosing groups
  Placebo: Placebo administered intramuscularly
Period: Overall Study
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01 | 100 mg of G03-52-01 | Pooled Placebo
Started | 7 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01 | 100 mg of G03-52-01 | Pooled Placebo | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.58) | 33.9 (6.69) | 35.8 (6.58) | 34 (4.04) | 36.3 (6.98) | 34.8 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 6 | 3 | 5 | 22
  Male | 3 | 4 | 2 | 5 | 3 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 7 | 4 | 5 | 24
  Not Hispanic or Latino | 3 | 4 | 1 | 4 | 3 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 7 | 8 | 6 | 7 | 33
  Other | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 75.77 (16.849) | 75.60 (13.001) | 74.59 (16.828) | 88.71 (12.486) | 87.15 (8.892) | 80.36 (13.611)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 27.47 (3.638) | 27.70 (4.419) | 28.44 (5.098) | 30.06 (1.907) | 31.03 (2.841) | 28.94 (3.58)
Height [Mean (Standard Deviation); unit: cm] | 165.39 (11.347) | 165.05 (5.190) | 161.45 (9.441) | 171.48 (10.268) | 167.86 (11.281) | 166.25 (9.51)

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of Serious Adverse Events (SAE) Following Administration of G03-52-01 to the Final Follow-up Visit.
Description: Determine number of SAEs after dosing (Cohorts 1-3)
Time Frame: day 0 to day 120
Measure: Number; unit: Number of SAEs
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01 | Pooled Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8
Number of SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: The Occurrence of Serious Adverse Events (SAE) Following Administration of G03-52-01 to the Final Follow-up Visit.
Description: Determine number of SAEs after dosing (Cohort 4)
Time Frame: day 0 to day 180
Measure: Number; unit: Number of SAEs
Arm/Group | 100 mg of G03-52-01 | Pooled Placebo
Number analyzed (Participants) | 8 | 8
Number of SAEs | 0 | 0

3. Primary Outcome: The Occurrence of Adverse Events (AE) Following Administration of G03-52-01 to the Final Follow-up Visit
Description: Determine number of AEs after dosing (Cohorts 1-3)
Time Frame: day 0 to day 120
Measure: Number; unit: Number of AEs
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01 | Pooled Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8
Number of AEs | 8 | 10 | 11 | 6

4. Primary Outcome: The Occurrence of Adverse Events (AE) Following Administration of G03-52-01 to the Final Follow-up Visit
Description: Determine number of AEs after dosing (Cohort 4)
Time Frame: day 0 to day 180
Measure: Number; unit: Number of AEs
Arm/Group | 100 mg of G03-52-01 | Pooled Placebo
Number analyzed (Participants) | 8 | 8
Number of AEs | 8 | 6

5. Primary Outcome: The Occurrence of Changes From Baseline in Physical Examination, Vital Signs and Clinical Safety Laboratory Values Following Administration of G03-52-01 to the Final Follow-up Visit.
Description: Determine number of changes from baseline (Cohorts 1-3)
Time Frame: day 0 to day 120
Measure: Number; unit: Number of events
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01 | Pooled Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8
Number of events | 7 | 3 | 7 | 4

6. Primary Outcome: The Occurrence of Changes From Baseline in Physical Examination, Vital Signs and Clinical Safety Laboratory Values Following Administration of G03-52-01 to the Final Follow-up Visit.
Description: Determine number of changes from baseline (Cohort 4)
Time Frame: day 0 to day 180
Measure: Number; unit: Number of events
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
Number of events | 1

7. Secondary Outcome: Serotype A Peak Plasma Concentration (Cmax)
Description: MNA assessment of PD (Cohorts 1-3)
Time Frame: pre-dose, days 4, 30, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
U/L | 0.0977 (46.37) | 0.288 (47.14) | 0.658 (49.29)

8. Secondary Outcome: Serotype A Peak Plasma Concentration (Cmax)
Description: MNA assessment of PD (Cohort 4)
Time Frame: pre-dose, 2 hours post-dose, days 4, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
U/L | 2.07 (79.84)

9. Secondary Outcome: Serotype B Peak Plasma Concentration (Cmax)
Description: MNA assessment of PD (Cohorts 1-3)
Time Frame: pre-dose, days 4, 30, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
U/L | 0.630 (100.37) | 1.30 (53.38) | 2.25 (57.90)

10. Secondary Outcome: Serotype B Peak Plasma Concentration (Cmax)
Description: MNA assessment of PD (Cohort 4)
Time Frame: pre-dose, 2 hours post-dose, days 4, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
U/L | 3.63 (20.85)

11. Secondary Outcome: Serotype A Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: MNA assessment of PD (Cohorts 1-3)
Time Frame: pre-dose, days 4, 30, 60, 90, and 120
Measure: Median (Full Range); unit: hrs
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
hrs | 96 [96 to 96] | 95.89 [95.6 to 96.98] | 96 [95.42 to 97.13]

12. Secondary Outcome: Serotype A Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: MNA assessment of PD (Cohort 4)
Time Frame: pre-dose, 2 hours post-dose, days 4, 30, 45, 60, 90, and 120
Measure: Median (Full Range); unit: hrs
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
hrs | 95.76 [93.95 to 96.2]

13. Secondary Outcome: Serotype B Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: MNA assessment of PD (Cohorts 1-3)
Time Frame: pre-dose, days 4, 30, 60, 90, and 120
Measure: Median (Full Range); unit: hrs
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
hrs | 96 [96 to 1394.55] | 96.78 [95.77 to 1463.82] | 96.01 [95.42 to 744.03]

14. Secondary Outcome: Serotype B Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: MNA assessment of PD (Cohort 4)
Time Frame: pre-dose, 2 hours post-dose, days 4, 30, 45, 60, 90, and 120
Measure: Median (Full Range); unit: hrs
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
hrs | 95.88 [93.95 to 695.88]

15. Secondary Outcome: Serotype A Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: MNA assessment of PD (Cohorts 1-3)
Time Frame: pre-dose, days 4, 30, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*U/L
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
h*U/L | 23.530 (174.61) | 82.821 (189.37) | 281.393 (33.21)

16. Secondary Outcome: Serotype A Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: MNA assessment of PD (Cohort 4)
Time Frame: pre-dose, 2 hours post-dose, days 4, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*U/L
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
h*U/L | 1106.673 (57.81)

17. Secondary Outcome: Serotype B Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: MNA assessment of PD (Cohorts 1-3)
Time Frame: pre-dose, days 4, 30, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*U/L
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
h*U/L | 608.306 (49.6) | 1208.471 (53.63) | 1939.427 (40.93)

18. Secondary Outcome: Serotype B Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: MNA assessment of PD (Cohort 4)
Time Frame: pre-dose, 2 hours post-dose, days 4, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*U/L
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
h*U/L | 2940.815 (33.14)

19. Secondary Outcome: Anti-BoNT A Peak Plasma Concentration (Cmax)
Description: ELISA/ECLA assessment of PK (Cohorts 1-3)
Time Frame: pre-injection, 2, 4, 8, 24, 48, and 72 hours post injection, and on days 4, 8, 15, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 10 mg of G03-52-01: 8 subjects randomized to 10 mg of G03-52-01
  G03-52-01: G03-52-01 administered intramuscularly
- 25 mg of G03-52-01: 8 subjects randomized to 25 mg of G03-52-01
  G03-52-01: G03-52-01 administered intramuscularly
Arm/Group | 10 mg of G03-52-01 | 25 mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
ng/mL | 123.06 (17.66) | 362.845 (33.605) | 678.635 (44.12)

20. Secondary Outcome: Anti-BoNT A Peak Plasma Concentration (Cmax)
Description: ELISA/ECLA assessment of PK (Cohort 4)
Time Frame: pre-injection, 6 hours post injection, and on days 1, 2, 4, 8, 15, 30, 45, 60, 90, 120, and 180
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
ng/mL | 1372.08 (33.69)

21. Secondary Outcome: Anti-BoNT B Peak Plasma Concentration (Cmax)
Description: ELISA/ECLA assessment of PK (Cohort 4)
Time Frame: pre-injection, 6 hours post injection, and on days 1, 2, 4, 8, 15, 30, 45, 60, 90, 120, and 180
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
ng/mL | 1668.88 (26.73)

22. Secondary Outcome: Anti-BoNT B Peak Plasma Concentration (Cmax)
Description: ELISA/ECLA assessment of PK (Cohorts 1-3)
Time Frame: pre-injection, 2,4, 8, 24, 48, and 72 hours post injection, and on days 4, 8, 15, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
ng/mL | 133.49 (18.73) | 401.25 (30.44) | 722.73 (37.85)

23. Secondary Outcome: Anti-BoNT A Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: ELISA/ECLA assessment of PK (Cohorts 1-3)
Time Frame: pre-injection, 2, 4, 8, 24, 48, and 72 hours post injection, and on days 4, 8, 15, 30, 45, 60, 90, and 120
Measure: Median (Full Range); unit: hrs
Arm/Group | 10 mg of G03-52-01 | 25 mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
hrs | 84 [48 to 359.53] | 71.71 [47.73 to 359.95] | 71.34 [48.07 to 192.02]

24. Secondary Outcome: Anti-BoNT A Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: ELISA/ECLA assessment of PK (Cohort 4)
Time Frame: pre-injection, 6 hours post injection, and on days 1, 2, 4, 8, 15, 30, 45, 60, 90, 120, and 180
Measure: Median (Full Range); unit: hrs
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
hrs | 47.87 [24.18 to 96]

25. Secondary Outcome: Anti-BoNT B Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: ELISA/ECLA assessment of PK (Cohorts 1-3)
Time Frame: pre-injection, 2, 4, 8, 24, 48, and 72 hours post injection, and on days 4, 8, 15, 30, 45, 60, 90, and 120
Measure: Median (Full Range); unit: hrs
Arm/Group | 10 mg of G03-52-01 | 25 mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
hrs | 128 [48 to 192] | 107.83 [47.73 to 359.95] | 79.58 [24.18 to 192.12]

26. Secondary Outcome: Anti-BoNT B Time to Achieve Peak Concentration of the Drug After Administration (Tmax)
Description: ELISA/ECLA assessment of PK (Cohort 4)
Time Frame: pre-injection, 6 hours post injection, and on days 1, 2, 4, 8, 15, 30, 45, 60, 90, 120, and 180
Measure: Median (Full Range); unit: hrs
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
hrs | 72.59 [24.18 to 192.12]

27. Secondary Outcome: Anti-BoNT A Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: ELISA/ECLA assessment of PK (Cohorts 1-3)
Time Frame: pre-injection, 2, 4, 8, 24, 48, and 72 hours post injection, and on days 4, 8, 15, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 10 mg of G03-52-01 | 25 mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
h*ng/mL | 76121.9 (32.64) | 211066.2 (29.35) | 346965.1 (33.76)

28. Secondary Outcome: Anti-BoNT A Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: ELISA/ECLA assessment of PK (Cohort 4)
Time Frame: pre-injection, 6 hours post injection, and on days 1, 2, 4, 8, 15, 30, 45, 60, 90, 120, and 180
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
h*ng/mL | 598555.3 (77.05)

29. Secondary Outcome: Anti-BoNT B Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: ELISA/ECLA assessment of PK (Cohort 1-3)
Time Frame: pre-injection, 2, 4, 8, 24, 48, and 72 hours post injection and on days 4, 8, 15, 30, 45, 60, 90, and 120
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 10 mg of G03-52-01 | 25 mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
h*ng/mL | 120541.5 (30.55) | 338924.7 (28.11) | 530432.5 (29.64)

30. Secondary Outcome: Anti-BoNT B Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: ELISA/ECLA assessment of PK (Cohort 4)
Time Frame: pre-injection, 6 hours post injection, and on days 1, 2, 4, 8, 15, 30, 45, 60, 90, 120, and 180
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
h*ng/mL | 1259300 (30.16)

31. Secondary Outcome: Anti-drug Antibodies (ADA)
Description: To assess the number of participants with positive anti-drug antibody levels (Cohorts 1-3)
Time Frame: pre-dose, days 15, 30, 45, 60, 90, and 120
Measure: Count of Participants; unit: Participants
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01
Number analyzed (Participants) | 7 | 8 | 8
Participants | 5 | 6 | 4

32. Secondary Outcome: Anti-drug Antibodies (ADA)
Description: To assess the number of participants with positive anti-drug antibody levels (Cohort 4)
Time Frame: pre-dose, days 45, 60, 90, 120, and 180
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg of G03-52-01
Number analyzed (Participants) | 8
Participants | 5

ADVERSE EVENTS:
Time Frame: 120 days for Cohorts 1-3 and 180 days for Cohort 4
Arm/Group | 10mg of G03-52-01 | 25mg of G03-52-01 | 50 mg of G03-52-01 | 100 mg of G03-52-01 | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/7 | 6/8 | 5/8 | 4/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10mg of G03-52-01 (N=7) | 25mg of G03-52-01 (N=8) | 50 mg of G03-52-01 (N=8) | 100 mg of G03-52-01 (N=8) | Pooled Placebo (N=8)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limbs stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Light headedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT04171115/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04171115/SAP_001.pdf